CLINICAL TRIAL: NCT04394741
Title: Effects of Dry Needling on Stiffness in Latent Myofascial Trigger Points: a Randomized Controlled Trial
Brief Title: Effects of Dry Needling on Stiffness in Latent Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNStiffness
Record Dates: First submitted 2020-05-10; First posted 2020-05-19 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Trigger Points
Keywords: Pain; Latent trigger point; Stiffness; Dry Needling
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Dry Needling (Experimental): Intervention-Dry Needling: Deep Dry Needing into the latent trigger point of the upper trapezius muscle
  Interventions: Device: Intervention-Dry Needling
- Sham Dry Needling (Sham Comparator): Control-Dry Needling: Sham Dry Needling into the latent trigger point of the upper trapezius muscle
  Interventions: Device: Intervention-Dry Needling; Device: Control-Dry Needling

INTERVENTIONS:
Device: Intervention-Dry Needling — Deep Dry Needling into the site of the latent Trigger Point of the upper trapezius muscle.
  1 session in upper trapezius muscle moving the needle up and down ten times.
Device: Control-Dry Needling — Sham Dry Needling into the site of the latent Trigger Point of the upper trapezius muscle with non-penetrating needles
  1 session in upper trapezius muscle moving the needle up and down ten times.
  Arms: Sham Dry Needling

SUMMARY:
The purpose of this study is to determine whether application of Dry Needling (DN) is effective for reduced on Stiffness in Latent trigger point (LTrP) of upper trapezius. The secondary purposes are to determine the correlation on two elastography for stiffness measure (Shear-wave elastography and Strain elastography). Randomized controlled trial, in parallel with cross-control design. Two groups with LTrP in upper trapezius, and will be randomly selected to DN group or Sham-Dn group.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30 years
* The presence of LTrP in the middle third of the upper trapezius muscle on the dominant side
* Being able to provide written informed consent
* Being able to follow instructions and realize clinical tests

Exclusion Criteria:

* Any pharmacological therapeutic
* Any medical treatment or physical therapies at cervical region during the 6-month before this study - Any diagnosed health problem
* Any history of head and upper extremity surgery or trauma
* Any red flags to DN, (ie: metabolic diseases, pregnancy, kinesiophobia, Infection, cancer)
* Absence of recurrent history of neck pain
* No neck pain symptomatology the previous 6 months
* Cervical disk herniation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change on Stiffness (Shear wave elastography and Strain Elastography) | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  Shear-wave Elastography (SWE) as assessed using an Logiq S8 US system (GE Healthcare).
  The stiffness was determined with measuring velocity of shear waves in trapezius muscle on SWE exam.
  Strain elastography (SEL) as assessed using an Logiq S8 US system (GE Healthcare).
  The stiffness was determined by applying light repetitive compression with the hand-held transducer

SECONDARY OUTCOMES:
Change in Pain Pressure Threshold (PPT) | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  Pressure-Pain Threshold as assessed by an manual mechanical algometer. PPT is the minimal amount of pressure that produces pain and is used to assess abnormalities in nociceptive processing or hyperalgesia.
Change in Thickness of muscle | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  The muscle was scanned in the longitudinal and axial planes, taking care to avoid anisotropy. B-Mode gray scale was employed to measure muscle thickness
Change in Post-needling soreness | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  The procedure performed was the subject had to characterize the level of pain using a visual analog scale (VAS), ranging from 0mm (no pain) to 10mm (worst imaginable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Abián-Vicén, PhD, Study Director — Castilla-La Mancha University
Locations (1):
- Performance and Sport Rehabilitation Laboratory, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruiz-Saez M, Fernandez-de-las-Penas C, Blanco CR, Martinez-Segura R, Garcia-Leon R. Changes in pressure pain sensitivity in latent myofascial trigger points in the upper trapezius muscle after a cervical spine manipulation in pain-free subjects. J Manipulative Physiol Ther. 2007 Oct;30(8):578-83. doi: 10.1016/j.jmpt.2007.07.014. PMID 17996549
- [Background] Grabowski PJ, Slane LC, Thelen DG, Obermire T, Lee KS. Evidence of Generalized Muscle Stiffness in the Presence of Latent Trigger Points Within Infraspinatus. Arch Phys Med Rehabil. 2018 Nov;99(11):2257-2262. doi: 10.1016/j.apmr.2018.03.024. Epub 2018 Apr 28. PMID 29709524
- [Background] Maher RM, Hayes DM, Shinohara M. Quantification of dry needling and posture effects on myofascial trigger points using ultrasound shear-wave elastography. Arch Phys Med Rehabil. 2013 Nov;94(11):2146-50. doi: 10.1016/j.apmr.2013.04.021. Epub 2013 May 14. PMID 23684553
- [Background] Luan S, Zhu ZM, Ruan JL, Lin CN, Ke SJ, Xin WJ, Liu CC, Wu SL, Ma C. Randomized Trial on Comparison of the Efficacy of Extracorporeal Shock Wave Therapy and Dry Needling in Myofascial Trigger Points. Am J Phys Med Rehabil. 2019 Aug;98(8):677-684. doi: 10.1097/PHM.0000000000001173. PMID 31318748
- [Derived] Sanchez-Infante J, Bravo-Sanchez A, Jimenez F, Abian-Vicen J. Effects of Dry Needling on Muscle Stiffness in Latent Myofascial Trigger Points: A Randomized Controlled Trial. J Pain. 2021 Jul;22(7):817-825. doi: 10.1016/j.jpain.2021.02.004. Epub 2021 Feb 23. PMID 33636373